CLINICAL TRIAL: NCT01338311
Title: Salbutamol: Tolerance to Bronchoprotection vs. Methacholine: Time Course of Onset
Brief Title: Salbutamol Tolerance Onset
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BMC 10-226
Record Dates: First submitted 2011-04-01; First posted 2011-04-19 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- salbutamol (Active Comparator)
  Interventions: Drug: salbutamol
- placebo (Placebo Comparator): 200mcg twice daily for a total of 7 doses
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: salbutamol — 200mcg twice daily for a total of 7 doses
  Arms: salbutamol
Drug: Placebo — 200mcg twice a day for a total of 7 doses (3.5 days).
  Arms: placebo

SUMMARY:
Overuse of inhaled bronchodilator beta agonist medication results in a loss of effectiveness (i.e. tolerance). This has been shown for the short acting beta agonist salbutamol and the long acting beta agonist salmeterol. Tolerance to salmeterol is present within 24 hours. The onset of tolerance to salbutamol is not known.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* 18 to 65 years of age
* non smoker
* beta agonist naive for at least 14 days
* baseline FEV1 at least 70% predicted
* no respiratory tract infection or allergen exposure (if atopic) within 4 weeks of visit 1

Exclusion Criteria:

* poorly controlled asthma
* pregnant or lactating women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Airway responsiveness as a measure of salbutamol bronchoprotection | ten minutes post 200mcg salbutamol on day 1
  Regular use of salbutamol results in loss of bronchoprotection. The primary outcome is to determine the onset of this tolerance.
Airway responsiveness as a measure of salbutamol bronchoprotection | ten minutes post 200mcg salbutamol on day 3
  Regular use of salbutamol results in loss of bronchoprotection. The primary outcome is to determine the onset of this tolerance.
Airway responsiveness as a measure of bronchoprotection. The primary outcome is to determine the onset of this tolerance. | ten minutes post 200mcg salbutamol on day 5
  Regular use of salbutamol results in loss of bronchoprotection. The primary outcome is to determine the onset of this tolerance.
Airway responsiveness as a measure of salbutamol bronchoprotection | ten minutes post 200mcg salbutamol on day 7
  Regular use of salbutamol results in loss of bronchoprotection. The primary outcome is to determine the onset of this tolerance.

CONTACTS AND LOCATIONS:
Overall Officials: Donald W Cockcroft, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Derived] Stewart SL, Martin AL, Davis BE, Cockcroft DW. Salbutamol tolerance to bronchoprotection: course of onset. Ann Allergy Asthma Immunol. 2012 Dec;109(6):454-7. doi: 10.1016/j.anai.2012.08.003. Epub 2012 Aug 22. PMID 23176887